CLINICAL TRIAL: NCT02132117
Title: Safety and Efficacy of Oxymetazoline HCl Cream 1.0% in Patients With Persistent Erythema Associated With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199201-005
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Results first posted 2016-08-02 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Erythema; Rosacea
MeSH Terms: conditions — Erythema; Rosacea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxymetazoline HCL Cream 1.0% (Experimental): Oxymetazoline HCL Cream 1.0% applied to the face once daily for 29 days.
  Interventions: Drug: Oxymetazoline HCL Cream 1.0%
- Vehicle (Placebo Comparator): Vehicle to Oxymetazoline HCL Cream applied to the face once daily for 29 days.
  Interventions: Drug: Vehicle to Oxymetazoline HCL Cream

INTERVENTIONS:
Drug: Oxymetazoline HCL Cream 1.0% — Oxymetazoline HCL Cream 1.0% (AGN-199201) applied to the face once daily for 29 days.
  Arms: Oxymetazoline HCL Cream 1.0%
Drug: Vehicle to Oxymetazoline HCL Cream — Vehicle to Oxymetazoline HCL Cream (AGN-199201) applied to the face once daily for 29 days.
  Arms: Vehicle

SUMMARY:
This study will evaluate the safety and efficacy of oxymetazoline hydrochloride (HCl) cream 1.0% (AGN-199201) once daily compared to vehicle for the treatment of persistent moderate to severe facial erythema associated with rosacea.

ELIGIBILITY:
Inclusion Criteria:

-Moderate to severe persistent facial erythema associated with rosacea.

Exclusion Criteria:

* Greater than 3 inflammatory lesions on the face
* Current treatment with monoamine oxidase (MAO) inhibitors
* Raynaud's syndrome, narrow angle glaucoma, orthostatic hypotension, scleroderma or Sjogren's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2014-06; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- College Station, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxymetazoline HCL Cream 1.0%: Oxymetazoline hydrochloride (HCL) Cream 1.0% applied to the face once daily for 29 days.
Period: Overall Study
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle
Started | 224 | 221
Completed | 213 | 216
Not Completed | 11 | 5
Not completed — Adverse Event | 6 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Personal Reasons | 1 | 2
Not completed — Other Miscellaneous Reasons | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle | Total
Number analyzed (Participants) | 224 | 221 | 445
Age, Customized [Number; unit: participants]
  18-64 years | 198 | 193 | 391
  >=65 years | 26 | 28 | 54
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 173 | 350
  Male | 47 | 48 | 95

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With at Least a 2-Grade Improvement (Decrease) From Baseline on Both Clinician Erythema Assessment (CEA) and Subject Self-Assessment for Rosacea Facial Redness (SSA) 5-point Scales
Description: The investigator assessed the participant's overall severity of erythema in the treatment area by using the 5-point CEA scale with photonumeric guide where: 0=clear skin with no signs of erythema (best) to 4=severe erythema; fiery redness (worst). A decrease in the score indicates improvement. The participant assessed their overall severity of rosacea facial redness in the treatment area by using the 5-point SSA scale with photoguide where: 0=no signs of unwanted redness (best) to 4=severe redness (worst). A decrease in the score indicates improvement. The percentage of participants with at least a 2-grade decrease (improvement) on both CEA and SSA from Baseline was evaluated over the 12-hour evaluation period (hours 3, 6, 9, and 12) post-dose on Day 29. Baseline was defined as the measurement at pre-dose on Day 1.
Time Frame: Baseline, Day 29 (Hours 3, 6, 9 and 12)
Population: Intent-to-treat (ITT) Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle
Number analyzed (Participants) | 224 | 221
percentage of participants
  Day 29 (Hour 3) | 14.3 | 7.4
  Day 29 (Hour 6) | 13.4 | 4.8
  Day 29 (Hour 9) | 15.5 | 8.5
  Day 29 (Hour 12) | 12.3 | 6.1

2. Secondary Outcome: Percentage of Participants With at Least a 2-Grade Improvement (Decrease) From Baseline on SSA at Hours 3, 6, 9 and 12 on Day 29
Description: The participant assessed their overall severity of rosacea facial redness in the treatment area by using the 5-point SSA scale with photoguide where: 0=no signs of unwanted redness (best) to 4=severe redness (worst). A decrease in the score indicates improvement. The percentage of participants with at least a 2-grade decrease (improvement) on SSA from Baseline was evaluated over the 12-hour evaluation period (hours 3, 6, 9, and 12) post-dose on Day 29.
Time Frame: Baseline, Day 29 (Hours 3, 6, 9 and 12)
Population: ITT Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle
Number analyzed (Participants) | 224 | 221
percentage of participants
  Day 29 (Hour 3) | 24.1 | 15.8
  Day 29 (Hour 6) | 24.8 | 14.7
  Day 29 (Hour 9) | 22.0 | 16.0
  Day 29 (Hour 12) | 23.7 | 15.8

3. Secondary Outcome: Percent Change From Baseline on Rosacea Facial Redness as Measured by Digital Imaging Analysis (DIA) at Hours 3, 6, 9 and 12 on Day 29
Description: DIA of photographs was used to assess rosacea facial redness and was defined as percentage of facial area occupied by redness. A higher value in the percentage of facial area occupied by facial redness indicated more redness. A negative/ lower number percent change from Baseline indicates improvement.
Time Frame: Baseline, Day 29 (Hours 3, 6, 9 and 12)
Population: ITT Population included all randomized participants.
Measure: Median (Full Range); unit: percent change in area of redness
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle
Number analyzed (Participants) | 224 | 221
percent change in area of redness
  Day 29 (Hour 3) | -25.70 (144.776) [-100.0 to 1666.0] | 0.00 (225.452) [-94.1 to 2864.7]
  Day 29 (Hour 6) | -15.95 (170.735) [-100.0 to 1760.3] | 2.25 (198.138) [-92.3 to 2037.4]
  Day 29 (Hour 9) | -10.95 (131.933) [-100.0 to 1067.2] | 5.15 (200.530) [-89.4 to 2037.4]
  Day 29 (Hour 12) | -9.60 (145.898) [-100.0 to 1486.9] | 1.00 (195.291) [-96.3 to 2037.4]

4. Secondary Outcome: Percentage of Participants Satisfied or Very Satisfied on Item #9 of Satisfaction Assessment for Rosacea Facial Redness (SAT-RFR) at Hours 3, 6, 9 and 12 on Day 29
Description: Participants assessed their treatment satisfaction by answering Item #9 of the SAT-RFR: "Right now, how satisfied are you with the effect your study medication had on your facial redness?" using a 5-point scale where 0= very dissatisfied, 1=dissatisfied, 2=neither satisfied or dissatisfied, 3=satisfied, or 4=very satisfied. The percentage of participants who answered Satisfied or Very Satisfied is reported.
Time Frame: Day 29 (Hours 3, 6, 9 and 12)
Population: Participants from the ITT Population, all randomized participants with data available for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle
Number analyzed (Participants) | 223 | 220
percentage of participants
  Day 29 (Hour 3) | 54.3 | 34.1
  Day 29 (Hour 6) | 49.3 | 32.3
  Day 29 (Hour 9) | 49.8 | 33.6
  Day 29 (Hour 12) | 47.5 | 36.4

5. Secondary Outcome: Change From Baseline on the Symptom Assessment for Rosacea Facial Redness (SA-RFR) Item # 4 at Hours 3, 6, 9 and 12 on Day 29
Description: Participants assessed the burning sensation associated with rosacea facial redness by answering Item #4 of the SA-RFR: "Right now, how much does your face burn because of your facial redness?" using a 5-point scale where 0=less severe to 4=severe. A negative change from Baseline indicates improvement.
Time Frame: Baseline, Day 29 (Hours 3, 6, 9 and 12)
Population: Participants from the ITT Population, all randomized participants, with data available for analysis at the given time-point. Only participants who had a SA-RFR score of 1-4 at Baseline are included in the Analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle
Number analyzed (Participants) | 129 | 134
score on a scale
  Day 29 (Hour 3) | -1.8 (0.97) | -1.6 (0.93)
  Day 29 (Hour 6) | -1.8 (0.93) | -1.6 (0.91)
  Day 29 (Hour 9) | -1.8 (0.91) | -1.7 (0.96)
  Day 29 (Hour 12) | -1.8 (0.92) | -1.7 (0.91)

6. Secondary Outcome: Percentage of Participants With at Least a 1-Grade Improvement (Decrease) From Baseline on SSA at Hour 1 on Day 1
Description: The participant assessed their overall severity of rosacea facial redness in the treatment area by using the 5-point SSA scale with photoguide where: 0=no signs of unwanted redness (best) to 4=severe redness (worst). A decrease in the score indicates improvement.
Time Frame: Baseline, Day 1 (Hour 1)
Population: ITT Population included all randomized participants.
Measure: Number; unit: percentage of participants
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle
Number analyzed (Participants) | 224 | 221
percentage of participants | 29.7 | 16.8

ADVERSE EVENTS:
Description: Safety Population, all participants who applied at least one dose of study medication, was used to determine the number of participants at risk for Serious Adverse Events and Adverse Events.
Arm/Group | Oxymetazoline HCL Cream 1.0% | Vehicle
Serious Adverse Events (participants affected / at risk) | 3/223 | 2/221
Other Adverse Events (participants affected / at risk) | 0/223 | 0/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxymetazoline HCL Cream 1.0% (N=223) | Vehicle (N=221)
Goitre (Endocrine disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Traumatic liver injury (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.